CLINICAL TRIAL: NCT03911492
Title: Canadian-American Spinal Cord Perfusion Pressure and Biomarker Study
Acronym: CASPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Rick Hansen Institute (Other)
Responsible Party: Principal Investigator, Brian Kwon, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-00805
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Acute Spinal Cord Injury; Acute Spinal Paralysis; Spinal Cord Injuries; SPINAL Fracture
Keywords: SCI; Spinal Cord Injury; CSF; Biomarker; CSF pressure; Traumatic SCI; Perfusion pressure
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCP Pressure Management (Other): Active management of Spinal Cord Perfusion Pressure (SCPP) at or above 65 mmHg.
  Interventions: Procedure: SCPP Management => 65 mmHg

INTERVENTIONS:
Procedure: SCPP Management => 65 mmHg — A lumbar intrathecal catheter will be inserted pre-operatively for the measurement of Intrathecal pressure (ITP) and the collection of cerebrospinal fluid (CSF) samples. SCPP will be calculated as the difference between Mean Arterial Pressure (MAP) and the ITP.

SUMMARY:
This multicenter study will enroll 100 patients with acute traumatic cervical and thoracic SCI who have a lumbar intrathecal catheter inserted within 24 hours of their injury. The lumbar intrathecal catheter will be inserted pre-operatively for the measurement of ITP and the collection of cerebrospinal fluid (CSF) samples. SCPP will be calculated as the difference between MAP and the ITP.

There are two important distinct yet related objectives in this prospective interventional study.

1. Determine the effect of SCPP maintenance ≥ 65 mmHg in acute SCI on neurologic recovery as measured by ASIA Impairment Scale (AIS) grade conversion and motor score improvement.
2. Collect CSF and blood samples for the measurement of neurochemical biomarkers and storage for future biomarker discovery and validation studies.

DETAILED DESCRIPTION:
Objective 1. To determine if actively maintaining an SCPP of at least 65 mmHg with a combination of MAP augmentation and CSF drainage promotes better neurologic recovery than routine hemodynamic management that focuses solely on MAP augmentation.

Objective 2. To determine if actively maintaining an SCPP of at least 65 mmHg with a combination of MAP augmentation and CSF drainage will allow for a reduction in the usage of vasopressors in acute SCI.

Objective 3. To determine the feasibility of draining CSF to reduce ITP in the acute post-injury setting, when the cord may be swollen against the dura causing subarachnoid space occlusion at the injury site.

Objective 4. To determine if there are complications associated with the installation of the intrathecal catheter and drainage of CSF in the acute SCI patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 17 (or the provincial age of majority - depending on local REB guidelines)
* Complete (AIS A) or incomplete (AIS B, C) acute traumatic spinal cord injury.
* Bony spinal levels between C0 and T12 inclusive.
* Blunt (non-penetrating) spinal cord injury treated either surgically or non-surgically
* Lumbar intrathecal catheter to be inserted as part of clinical hemodynamic management and CSF sample collected within 48 hours of injury
* Initial blood sample collected within 24 hours of injury

Exclusion Criteria:

* Motor incomplete spinal cord injury AIS D (i.e. at least half (half or more) of the key muscle functions below the neurological level of injury (NLI) have a muscle grade greater than or equal to 3/5)
* Spinal cord injury with sensory deficit only (i.e. no motor deficit)
* Penetrating spinal cord injury (including gunshot wounds)
* Isolated radiculopathy
* Isolated cauda equina injury or spinal injury below L1
* Associated injury (soft tissue or bony) to the lumbar spine where the intrathecal catheter would be placed
* Associated traumatic conditions that would interfere with the outcome assessment (e.g., traumatic brain injury, chest, pelvis, abdomen, or femur injury requiring operative intervention)
* Pre-existing neurodegenerative disorder, such as Parkinson's disease, Alzheimer's disease, Huntington's disease, multiple sclerosis, amyotrophic lateral sclerosis
* Pre-existing thromboembolic disease or coagulopathy, such as hemophilia, von Willebrand disease
* Presence of systemic disease that might interfere with patient safety, compliance or evaluation of the condition under study (e.g., clinically significant cardiac disease, HIV, Hep B or C) HTLV-1
* Pre-existing inflammatory or autoimmune disorder (e.g. rheumatoid arthritis, systemic lupus, psoriasis, or ankylosing spondylitis
* Any other medical condition that in the investigator's opinion would render the protocol procedures dangerous or impair the ability of the patient to receive protocol therapy
* Female patients who are pregnant

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examination | 12 months
  Neurologic recovery over time will be measured using the ISNCSCI examination - at Baseline, Days 1-7, and months 3, 6 and 12. Our primary outcome measure will be the change in total motor score at 6 months post-injury (a time point at which most motor recovery has occurred and is commonly used in acute SCI clinical trials).

SECONDARY OUTCOMES:
Levels of specific biochemical markers in CSF and Blood | 7 days
  CSF and blood samples will be obtained from the intrathecal catheter at 8-hour intervals, three times daily, for 7 days. These samples will be markers that correlate with injury severity and predict neurological outcome.
Spinal Cord Perfusion Pressure (SCPP) | 7 days
  SCPP will be calculated as the difference between the mean arterial pressure and intrathecal pressure. The MAP and ITP will recorded over 7 days post injury.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kwon, MD, PhD, Principal Investigator — University of British Columbia, Faculty of Medicine
Locations (8):
- United States (4):
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Halifax Infirmary - QEII, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No